CLINICAL TRIAL: NCT05636085
Title: Clinical Performance of the Mainz Biomed Colorectal Cancer Screening Test for the Detection of Colorectal Cancer and Advanced Adenoma in an Average Risk Population
Brief Title: Clinical Performance of the Mainz Biomed Colorectal Cancer Screening Test for Colorectal Cancer and Advanced Adenoma
Acronym: reconAAsense
Status: Not yet recruiting | Type: Observational
Sponsor: Mainz Biomed (Industry)
Responsible Party: Sponsor
Other Study IDs: MNZ-CRC-001
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Polyp; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Eligible subjects: Subjects ≥45 years of age and at average risk of colorectal cancer.
  Interventions: Device: Mainz Biomed Colorectal Cancer Screening Test

INTERVENTIONS:
Device: Mainz Biomed Colorectal Cancer Screening Test — There is no intervention.

SUMMARY:
This study is to determine how the Mainz Biomed Colorectal Cancer Screening Test works when used in people aged ≥45 years of age and at an average risk of developing colorectal cancer.

DETAILED DESCRIPTION:
This study is to validate the clinical performance for the Mainz Biomed Colorectal Cancer Screening Test in an average risk population aged ≥45 years of age.

Stool samples will be collected from subjects ≥45 years of age, of average risk for colon cancer, and scheduled to have a screening colonoscopy. The samples will be collected prior to colonoscopy and will be tested with the Mainz Biomed Colorectal Cancer Screening Test. The results will be compared with colonoscopy results to determine test performance.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is any sex and ≥45 years of age
2. Subject must be advised to have or be scheduled for a screening colonoscopy
3. Subject is at average risk for colorectal cancer according to the United States Preventive Services Task Force (USPSTF) guidelines, including:

   * no prior diagnosis of colorectal cancer, adenomatous polyps, or inflammatory bowel disease
   * no personal diagnosis or family history of known genetic disorders that predispose them to a high lifetime risk of colorectal cancer including:

     * Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease
     * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP)
     * Hereditary non-polyposis colorectal cancer syndrome (also referred to as "HNPCC" or "Lynch Syndrome")
     * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardner's Syndrome, Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis and Familial Hyperplastic Polyposis
     * Cronkhite Canada Syndrome
4. Subject can understand the study procedures and is able to provide consent to participate in the study and authorizes release of relevant protected health information through reviewing and consenting to a Health Insurance Portability and Accountability Act (HIPAA) medical release form
5. Subject is able and willing to provide stool samples within ninety (90) days before the colonoscopy procedure
6. Subject is able and willing to undergo a colonoscopy after providing a stool sample

Exclusion Criteria:

1. Subject had any precancerous findings on most recent colonoscopy.
2. Subject has a history of abnormal imaging suggesting colorectal cancer (e.g., colonography, MRI, CT, barium enema)
3. Subject has a history of any of the following cancers: oral, head and neck, lung, esophagus, gastric, biliary/liver, pancreatic, small bowel, or appendiceal
4. Subject has had a positive non-invasive screening diagnostic within the associated recommended intervals

   * High-sensitivity fecal occult blood test or fecal immunochemical test within the previous twelve (12) months
   * sDNA-FIT test within the previous thirty-six (36) months
5. Subject has had a colonoscopy in the previous nine (9) years
6. Subject has had a prior colorectal resection for any reason other than sigmoid diverticular disease
7. Indication for colonoscopy due to overt rectal bleeding (e.g., hematochezia or melena) within the previous thirty (30) days
8. Subject has any condition that in the opinion of the investigator should preclude participation in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects that have been advised to have or are scheduled for a screening colonoscopy.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity Colorectal Cancer | 18 to 24 months
  Sensitivity of the Mainz Biomed Colorectal Cancer Screening Test for Colorectal Cancer
Sensitivity Advanced Adenoma | 18 to 24 months
  Sensitivity of the Mainz Biomed Colorectal Cancer Screening Test for Advanced Adenoma
Specificity | 18 to 24 months
  Specificity of the Mainz Biomed Colorectal Cancer Screening Test for Advanced Neoplasia

SECONDARY OUTCOMES:
Positive predictive value and negative predictive value | 18 to 24 months
  Determine the positive predictive value and negative predictive value for the Mainz Biomed Colorectal Cancer Screening Test for Colorectal Cancer, Advanced Adenoma, and Advanced Neoplasia

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kim Turgeon, MD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No